CLINICAL TRIAL: NCT01591954
Title: A Feasibility/Pilot Study of a Modular Video Augmentation System for Image-Guided Endoscopic Skull Base Surgery
Brief Title: A Feasibility Study of a Modular Video Augmentation System for Image-Guided Skull Base Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 3rd party proprietary software issue
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: J11101; NA_00051786 (Other: JHMIRB)
Record Dates: First submitted 2012-05-01; First posted 2012-05-04 (Estimated); Results first posted 2016-12-01 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-10

CONDITIONS: Feasibility of Video Augmentation System; Value of Video Augmentation Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Video Augmentation (Experimental): Qualitative assessment of the value of video-based navigation system
  Interventions: Device: Video Augmentation

INTERVENTIONS:
Device: Video Augmentation — Assessment of value of video-based navigation system
  Other Names: Interfaces with Medtronic Stealthstation

SUMMARY:
Current standard of care for complex head, neck and skull base surgery require navigation systems that allow instruments to be tracked optically or electromagnetically while registered to a patient's pre-operative X-ray computed tomography (CT) or magnetic resonance image (MRI). However, conventionally, the CT/MRI data is not registered with video endoscopy. Augmentation of endoscopic video by preoperative data can facilitate navigation around critical structures and robust target resection. The work presented here describes evaluation of a high definition (HD) video-overlay system for endonasal endoscopic skull base surgery. We adopt a modular design that can be extended for other video augmentation applications. The system supports fast automatic camera calibration, comparable in re-projection errors to standard camera calibration tools, while performing within appropriate run time for clinical use. Phantom studies have shown the registration accuracy of the system to be equivalent to that of conventional optical tracking. With this system we are proposing a clinical pilot study in a small number of patients at Johns Hopkins Hospital to evaluate basic feasibility and to gather qualitative assessment of the video augmentation system.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years of age or older;
* Have an existing clinically ordered CT image within 2 weeks of the study; or
* Have an existing clinically ordered MR image within 2 weeks of the study;
* Provide written informed consent after receiving a verbal and written explanation of the purpose and nature of this clinical study;
* Be able to communicate effectively with clinical study personnel

Exclusion Criteria:

* Major medical or psychiatric illness which, in the investigator's opinion, would prevent completion of the procedure;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary L Gallia, M.D., Ph.D., Principal Investigator — Johns Hopkins Hospital Department of Neurosurgery
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Video Augmentation
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Video Augmentation
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Qualitative Assessment of Video Augmentation Software by Post-operative Survey of Neurosurgeon and Otolaryngologist
Description: The qualitative assessment of new video augmentation software by the three surgeons surveys the effect of video augmentation overlay on overall surgical confidence, procedure, approach, and visualization.
  1. = Significant hindrance / Negative effect;
  2. = Minor hindrance / Slightly negative effect;
  3. = Not helpful / No benefit or hindrance;
  4. = Somewhat helpful / Slight benefit;
  5. = Very helpful / Major benefit. Evaluation of safety is determined by collecting data regarding additional time, personnel and possible contamination.
Time Frame: Assessment is immediate, following operation.
Population: The study was terminated following 1 subject accrual. The system encountered basic software incompatibility and would not function reliably. The problem could not be resolved even with extensive technical troubleshooting, so the study was terminated. Data was collected for one participant but could not be analyzed due to software incompatibility.
Arm/Group | Video Augmentation
Number analyzed (Participants) | 0

2. Secondary Outcome: Data Recording for Retrospective Analysis
Description: The secondary outcome variable of this study is the data recorded by the video augmentation system during pertinent portions of the operation. We will be targeting steps in the procedure that would have the greatest benefit from an augmented video scene to be used later for further studies. Such data will form the subject of retrospective analysis of workflow.
  Three sets of data will be collected to be able to reconstruct the video scene for analysis of the system:
  1. - Tracked Endoscope information.
  2. - Video from endoscopy
  3. - Planning CT/MRI data
Time Frame: Data is recorded during case.
Population: as for outcome 1
Arm/Group | Video Augmentation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Video Augmentation
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes